CLINICAL TRIAL: NCT02080286
Title: Boosting the Therapeutic Benefits of Prism Adaptation by Combining it With tDCS
Brief Title: Transcranial Stimulation (tDCS) and Prism Adaptation in Spatial Neglect Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 12/sc/0556
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Spatial Neglect; Stroke; Cerebrovascular Disorders; Cerebral Infarction; Brain Diseases
Keywords: spatial neglect; rehabilitation; brain stimulation; tDCS; prism adaptation
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Cerebral Infarction; Brain Diseases | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Prism adaptation + anodal tDCS (Active Comparator): Participants will receive 1 milliamp (mA) anodal tDCS over the left primary motor cortex concurrent with a 20-minute session of prism adaptation.
  They will undergo 5 consecutive daily sessions.
  Interventions: Behavioral: Prism Adaptation; Device: Anodal tDCS
- Prism Adaptation + Sham tDCS (Placebo Comparator): Participants will receive Sham tDCS over the left primary motor cortex concurrent with a 20-minute session of prism adaptation.
  They will undergo 5 consecutive daily sessions.
  Interventions: Behavioral: Prism Adaptation; Device: Sham tDCS
- Prism adaptation + no tDCS (Placebo Comparator): Participants will receive no tDCS at all but will undergo a 20-minute session of prism adaptation.
  They will undergo 5 consecutive daily sessions.
  Interventions: Behavioral: Prism Adaptation

INTERVENTIONS:
Behavioral: Prism Adaptation — All participants will undergo prism adaptation, a form of behavioural therapy involving reaching and pointing movements while wearing glasses that induce an optical shift.
Device: Anodal tDCS — Participants will receive 1mA anodal tDCS over the left primary motor cortex. The active (positive) electrode will be centered on the scalp overlying the primary motor cortex and the reference (negative) electrode will be placed over the contralateral supraorbital ridge.
  The stimulation will last 20 minutes and run concurrent with the duration of the prism adaptation therapy.
  Arms: Prism adaptation + anodal tDCS
Device: Sham tDCS — Participants will receive 1mA sham tDCS over the left primary motor cortex. The active (positive) electrode will be centered on the scalp overlying the primary motor cortex and the reference (negative) electrode will be placed over the contralateral supraorbital ridge.
  The stimulation will last 20 minutes and run concurrent with the duration of the prism adaptation therapy.
  Arms: Prism Adaptation + Sham tDCS

SUMMARY:
The present study aims to compare the relative therapeutic efficacy of prism adaptation therapy combined with real versus sham tDCS. The investigators will test the hypothesis that the magnitude and duration of neglect improvement will be increased when prism therapy is combined with real tDCS compared to sham tDCS.

A second objective is to test whether individual differences in baseline clinical or brain imaging measures can predict: 1) neglect severity or 2) inter-individual differences in patients' therapeutic response.

A third goal is to use brain imaging to characterize the patterns of neural change induced by the intervention to identify brain structures that mediate therapeutic response.

DETAILED DESCRIPTION:
'Neglect' is a common neurological syndrome that affects approximately 50% of right-hemisphere stroke patients. It is a complex multi-faceted syndrome, but its core defining feature is that patients lose the capacity to voluntarily control attention in the left half of space. Neglect has a significant debilitating effect on patients' functional independence and everyday life and indicates a poor prognosis for long-term functional recovery.

To date, there is no effective rehabilitation intervention available for routine clinical use. One of the most promising experimental strategies for neglect rehabilitation is prism adaptation, a form of motor training that induces short-lived improvements in a variety of cognitive domains. However, its major limitation is that the benefits are transient. The investigators aim to test the hypothesis that by combining prism therapy with transcranial direct current stimulation (tDCS), this will boost learning/memory processes, resulting in larger and longer-lasting therapeutic effects.

The investigators will conduct a randomized controlled clinical trial to test the efficacy of multi-session prism therapy combined with real versus sham tDCS for the rehabilitation of chronic post-stroke neglect. Baseline neuroimaging data will be used as predictor variables to explain inter-individual variation in therapeutic response. Contrasts between pre- and post-intervention imaging data will be performed to identify neural structures that mediate therapeutic effects.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18-85
* At least one month post ischaemic or haemorrhagic stroke or brain damage to the right hemisphere
* Diagnosis of neglect confirmed by evidence of neglect on at least one of the tests in the battery of neglect tests administered during the Recruitment Interview

Absolute contraindications to participation in any part of the study:

* Anyone who does not have adequate understanding of English, sufficient to give informed consent
* Limited verbal communication in the form of dysphasia
* Any person who has a history of drug abuse as the data collected may be influenced by their condition
* Any person who has a history of dementia or any other psychiatric illness as the data collected may be influenced by their condition

Absolute contraindications to participation in the tDCS part of the study:

* Anyone who has a previous personal history of epilepsy, seizures, febrile convulsions as a child or recurrent fainting fits will be excluded from the tDCS part of the study
* Any metallic implant in the neck, head, or eye that is situated within the path of the tDCS current, and anyone with any implanted electrical devices, would be excluded as there is a risk of heating with tDCS
* Pregnant women are excluded as a precaution as there are no data on the effect on maternal tDCS or MRI on the foetus

Absolute contraindications to participation in the MRI part of the study:

* People who suffer from claustrophobia will be excluded from the MRI part of the study if they state they are unable to tolerate the scanner environment
* Anyone with a metal implant or implantable device that is found to be unsafe or unknown for MRI following investigations by named researchers and staff radiographers would be excluded.
* Pregnant women are excluded as a precaution as there are no data on the effect on maternal tDCS or MRI on the foetus

Potential contraindications to participation in the tDCS part of the study:

* Participants on some prescription medications such as anti-depressants or pain medication may be excluded as they may be at an increased risk of seizure
* Individuals who have a family history of epilepsy or seizure may be excluded as this may increase the individual's personal risk of susceptibility to seizures

Potential contraindications to participation in the MRI part of the study:

• An individual with a previous history of a surgical procedure may be excluded, depending on whether a metallic implant was used in their operation and whether the MRI-safety status of the implanted materials can be adequately assessed after requesting the medical/surgical notes (with patient consent) and/or post-surgical imaging and consulting with the staff radiographers who are legally responsible for determining participant safety in advance of any scanning.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-02; Primary Completion 2018-05 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Behavioural Inattention Test (BIT) | Assessed at the recruitment interview (week 0) and at the exit interview (8 weeks after the intervention)
  Change in score between the baseline session and the late post-intervention session.
Neglect Test Battery | Assessed at 2 separate pre-intervention baseline sessions at least 1 week apart. Re-assessed following the intervention at intervals of 1, 2, 4 and 8 weeks.
  This battery features a range of computerized and paper-and-pencil tests of neglect (eg: cancellation, eye movement recordings, etc.). We are testing for the percentage change in performance on this battery from the baseline pre-intervention phase at each of the post-intervention timepoints.

SECONDARY OUTCOMES:
Changes in brain imaging data | Change in a range of MRI measures between one baseline pre-intervention scan and the post-intervention scan (+ 5 weeks)
  We will test for changes in a range of MRI measures which we expect to be induced by the therapeutic intervention (measures of resting state and task functional MRI signal, grey and white matter, brain chemistry).

CONTACTS AND LOCATIONS:
Overall Officials: Jacinta O'Shea, Dr, Principal Investigator — University of Oxford
Locations (1):
- FMRIB Centre, John Radcliffe Hospital, University of Oxford, Oxford, United Kingdom

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411